CLINICAL TRIAL: NCT03583710
Title: A Randomized Registry Trial of Adjuvant Mitotane vs. Mitotane With Cisplatin/Etoposide After Primary Surgical Resection of Localized Adrenocortical Carcinoma With High Risk of Recurrence (ADIUVO-2 Trial)
Brief Title: Mitotane With or Without Cisplatin and Etoposide After Surgery in Treating Patients With Stage I-III Adrenocortical Cancer With High Risk of Recurrence
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0948; NCI-2018-01101 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0948 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: ENSAT Stage I Adrenal Cortex Carcinoma; ENSAT Stage II Adrenal Cortex Carcinoma; ENSAT Stage III Adrenal Cortex Carcinoma
MeSH Terms: interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; Mitotane; Dichlorodiphenyldichloroethane; Ethane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm A (mitotane) (Experimental): Patients receive mitotane PO daily on days 1-21. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Mitotane; Other: Quality-of-Life Assessment
- Arm B (mitotane, etoposide, cisplatin) (Experimental): Patients receive mitotane as in Arm A. Patients also receive cisplatin IV over 2 hours on day 1 and etoposide IV over 2 hours on days 1-3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Etoposide; Drug: Mitotane; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm B (mitotane, etoposide, cisplatin)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
  Arms: Arm B (mitotane, etoposide, cisplatin)
Drug: Mitotane — Given PO
  Other Names: (o,p)-DDD; 1, 1-Dichloro-2-(o-chlorophenyl)-2-(p-chlorophenyl)ethane; 1-Chloro-2-[2,2-dichloro-1-(4-chlorophenyl)ethyl]benzene; 2, 2-Bis(2-chlorophenyl-4-chlorophenyl)-1,1-dichloroethane; 2, 4''-Dichlorodiphenyldichloroethane; CB 313; CB-313; Chloditan; Chlodithane; DDD; Ethane, 2-(o-chlorophenyl)-2-(p-chlorophenyl)-1,1-dichloro-; Khloditan; Lisodren; Lysodren; Mytotan; o,p'' - DDD; o,p''-DDD; Ortho,para-DDD; WR-13045
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase III trial studies how well mitotane alone works compared to mitotane with cisplatin and etoposide when given after surgery in treating patients with adrenocortical cancer that has a high risk of coming back (recurrence). Cortisol can cause the growth of adrenocortical tumor cells. Antihormone therapy, such as mitotane, may lessen the amount of cortisol made by the body. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether mitotane alone or mitotane with cisplatin and etoposide after surgery works better in treating patients with adrenocortical carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the effect of adjuvant mitotane treatment alone (arm A) with that of adjuvant mitotane combined with four 21-day cycles of etoposide/cisplatin (arm B) on recurrence-free survival (RFS) in patients with high-risk adrenocortical carcinoma (ACC) after initial surgical resection.

SECONDARY OBJECTIVES:

I. Assess overall survival (OS), defined as the time interval between the date of randomization and the date of death from any cause.

II. Assess the effect of serum mitotane levels, disease stage, and surgical resection margins on clinical outcomes.

III. Assess the effect of early start (1-6 weeks from surgery) versus (vs.) late start (> 6 weeks from surgery) of adjuvant therapy on clinical outcomes.

IV. Assess serious adverse events. V. Measure quality of life at baseline, 6 weeks, 6 months after the initiation of adjuvant therapy, and at the end of study participation (recurrence or completing study treatments) using a validated quality of life questionnaire (European Organization for Research and Treatment of Cancer [EORTC] QLQ-C30).

EXPLORATORY OBJECTIVES:

I. Perform molecular profiling on available tissue specimens obtained at the time of initial surgical resection (formalin-fixed paraffin-embedded or frozen tissues) to identify genomic alterations in primary tumors that are associated with the clinical end points.

II. Evaluate markers to detect ACC recurrence or predict response to therapy (including steroid hormones and precursors, circulating tumor cells, and micro ribonucleic acid [microRNA]).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive mitotane orally (PO) daily on days 1-21. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive mitotane as in Arm A. Patients also receive cisplatin intravenously (IV) over 2 hours on day 1 and etoposide IV over 2 hours on days 1-3. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of ACC (Weiss score of >= 3). (LinWeiss-Bisceglia system will be used for oncocytic ACC).
* Have a high risk of relapse defined as: Stage I-III ACC (according to the European Network for the Study of Adrenal Tumors [ENSAT] classification) within 90 days of surgical resection of primary tumor with curative intent with either microscopically complete resection (R0, defined as no evidence of microscopic residual disease according to surgical reports, histopathology, and perioperative imaging), microscopically positive margins (R1), or undetermined margins (RX, based on surgical or pathological reports without unequivocal evidence of metastasis in the perioperative imaging). Each participating center will determine the pathological stages and resection margins AND Ki67 > 10% (to be determined by an experienced pathologist in each participating center and preferably via quantitative imaging analysis).
* Have perioperative imaging (computed tomography [CT] with contrast, magnetic resonance imaging [MRI] of the chest/abdomen/pelvis, or fluorodeoxyglucose positron emission tomography [FDG-PET] CT) without unequivocal evidence of disease within 8 weeks before randomization. Patients with indeterminate non-specific nodules (< 1 cm for soft tissue lesions and < 1.5 cm in the short dimension for lymph nodes) will be permitted to participate in this study.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Be able to comply with the protocol procedures.
* Provide written informed consent.

Exclusion Criteria:

* The time between primary surgery and randomization > 90 days.
* Gross residual disease after surgery (R2 resection)
* High suspicion for metastatic disease on perioperative imaging
* They have undergone repeated surgery for recurrence of disease.
* They have a history of recent or active prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, breast ductal carcinoma in situ, or other treated malignancies where there has been no evidence of disease for at least 2 years.
* They have renal insufficiency (estimated glomerular filtration rate [GFR] < 50 mL/min/1.73 m^2).
* They have significant liver insufficiency (serum bilirubin > 2 times the upper normal range)
* They have significant liver insufficiency (serum alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 3 times the upper normal range)
* Impaired bone marrow reserve (neutrophils < 1000/mm^3)
* Impaired bone marrow reserve (platelets < 100,000/mm^3)
* Pregnancy or breast feeding.
* They have known congestive heart failure (ejection fraction < 45%). The extent of cardiac testing will depend on the judgment of the local principal investigator (PI). In general, in patients with a history of cardiac disease, it is recommended to obtain a baseline two-dimensional echocardiogram as standard of care to document ejection fraction. In patients without prior cardiac disease, a baseline electrocardiogram (EKG) is sufficient if there is no evidence of acute ischemic changes or prior evidence of myocardial infarction. If EKG results are abnormal (ischemic changes, significant arrhythmia, or suggestion of prior myocardial infarction), a two-dimensional echocardiogram will be obtained to assess ejection fraction. Cardiac imaging and EKG may not be needed in patients assigned to mitotane who do not have prior cardiac history and have low suspicion for cardiac symptoms to reflect standards of clinical practice. Similarly, utilizing cardiac imaging and EKG within the past 12 months is permitted if there is no suspicion for cardiac issues.
* They have preexisting grade 2 peripheral neuropathy.
* They underwent previous or current treatment with mitotane or other antineoplastic drugs for ACC.
* They underwent previous radiotherapy for ACC.
* They have any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would, in the judgment of the investigator, pose excess risk associated with study participation or administration of the involved drugs or that, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | From the time of randomization up to 2 years
  Starting from the date of randomization until documentation of radiological evidence of local recurrence, radiological evidence of distant recurrence, or death from any cause (whichever occurs first), RFS will be compared using the log-rank test between the two arms.
Local recurrence of adrenocortical carcinoma (ACC) | Up to 6 months
Distant recurrence of ACC | Up to 6 months

SECONDARY OUTCOMES:
Overall survival (OS) | From the time of randomization up to 2 years
  Overall survival will be compared using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Jeena Varghese, Principal Investigator — M.D. Anderson Cancer Center
Locations (23):
- United States (3):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - M D Anderson Cancer Center, Houston, Texas
- France (16):
  - Institut de Cancérologie de l'Ouest (ICO), Angers
  - CHU Angers, Hôpital Larrey, Angers
  - CHU Besançon, Hôpital Jean Minjoz, Besançon
  - CHU Brest, Hôpital La Cavale Blanche, Brest
  - Centre Georges François Leclerc, Dijon
  - HCL Hôpital Louis Pradel, Lyon
  - CHU Nantes, Hôpital René et Guillaume Laënnec, Nantes
  - Hôpital Cochin, AP-HP, Paris
  - CHU Bordeaux - Hôpital Haut Lévèque, Pessac
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - HUS, Hôpital Hautepierre, Strasbourg
  - ICANS Institut de cancérologie Strasbourg Europe, Strasbourg
  - CHU Toulouse, Hôpital Larrey, Toulouse
  - CHU Toulouse, Hôpital Rangueil, Toulouse
  - Gustave Roussy, Villejuif
- Maria Sklodowska-Curie National Research Institute of Oncology, Gliwice, Poland
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
  - Akademiska Sjukhuset, Uppsala

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org